CLINICAL TRIAL: NCT05488795
Title: Identifying Successful Strategies for Implementing Team-Based Home Blood Pressure Monitoring in Primary Care
Brief Title: Team-Based Home Blood Pressure Monitoring
Acronym: TB-HBPM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kevin Fiscella, Professor, Family Medicine, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: RSRB 6036; R33HL157643 (NIH)
Record Dates: First submitted 2022-07-06; First posted 2022-08-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: High Blood Pressure; Hypertension
Keywords: Home blood pressure monitoring; Hypertension control; Primary Care Teams; Implementation Research; Health Equity; Clinical Trial
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Cluster Randomized Design. Each practice suite represents a cluster. All eight suites begin in the control group and then cross over (one-way) to the intervention group at one of three randomly assigned time periods, ensuring that all suites eventually receive implementation of TB-HBPM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Suite TB-HBPM pre intervention (Other): Each suite/cluster throughout the institution will begin in the baseline usual care phase in the first year.
  Interventions: Behavioral: Team-Based Home Blood Pressure Monitoring
- Suite TB-HBPM throughout intervention implementation (Other): Each suite will be randomized to implement the TB-HBPM program during one of three wedges separated by six months between each, 1.5 years later.
  Interventions: Behavioral: Team-Based Home Blood Pressure Monitoring
- Suite TB-HBPM post intervention implementation (Other): Post implementation phase of the suites 2 years after introduction of intervention.
  Interventions: Behavioral: Team-Based Home Blood Pressure Monitoring

INTERVENTIONS:
Behavioral: Team-Based Home Blood Pressure Monitoring — Implementation of best practices for hypertension control using a practice wide team-based home blood pressure monitoring intervention

SUMMARY:
The overall goal of this study is to identify and rigorously evaluate strategies for implementing and sustaining team-based home blood pressure monitoring (TB-HBPM) within primary care.

The TB-HBPM intervention is a multifaceted program involving patient transmission of blood readings to EHR and clinical decision support. Implementation strategies include group-based education on hypertension measurement, target blood pressure goals, drug and lifestyle management, referral to community resources, and team training designed to optimize the coordination of hypertension care, and monthly audit and feedback reports to teams and clinicians.

Hypertension control rates are suboptimal in many primary care practices with persistent racial disparities in control. Team-based home blood pressure monitoring (TB-HPBM) involving patient transmission of their home blood pressure readings in real-time to their clinical team has been shown to improve blood pressure control. There is an urgent need to implement TB-HBPM into practice. The overall objective of this research is to assess implementation strategies that mitigate barriers and leverage facilitators to TB-HBHM on hypertension control and disparities between Black and White patients. The study team and investigators will use mixed methods to assess the process and generate knowledge to facilitate broader uptake of TB-HBPM.

DETAILED DESCRIPTION:
Aim 2: Deploy theorized implementation strategies using a type-2 hybrid stepped-wedge randomized cluster trial The department of family medicine will roll out the clinical intervention (TBHBPM).

To improve rigor in evaluation, the study biostatistician will use computer-generated numbers to randomly assign each of the eight suites to when they will begin the intervention during one of three wedges (Figure 1). The study team and investigators will randomize two suites in the first wedge and three each to the second and third wedge.

Aim 3: Assess the impact of implementation strategies using specific metrics based on RE-AIM

Aim 4: Test theoretical assumptions underlying the implementation strategies

ELIGIBILITY:
ELIGIBILITY CRITERIA

Clinicians and Staff Eligibility Criteria Practice employees (practice leaders, administrators, clinicians, or staff) that work with hypertensive patients during the study period (scheduling appointments, coordinating care, measuring blood pressure, responding to questions, and/or treating their blood pressure)

Patient Inclusion Criteria

* Current HFM patient 18-85 years of age with hypertension diagnosis
* Diagnosis of hypertension based on ICD-10 codes of I10-I14
* at least one HFM health visit and hypertension diagnosis beginning no later than 7/1/2021.

Patient Exclusion Criteria

* Not current patient in the participating practices
* Diagnosis of dementia, end-stage renal disease, and/or in hospice
* Currently pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5760 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure control | Up to 48 months participation
  Change in percent of participants whose BP is controlled (defined as <140/90 mm Hg) among all eligible patients diagnosed with hypertension based on the last BP reading during the control period and the last BP reading during the follow-up period.

SECONDARY OUTCOMES:
Blood pressure control by race and ethnicity | Up to 48 months participation
  Change in percent of participants with blood pressure controlled defined as <140/90 mm Hg by race/ethnicity: among eligible Non-Hispanic White patients, non-Hispanic Black patients, and Hispanic patients.
Blood pressure control by insurance | Up to 48 months participation
  Change in percent of participants with blood pressure controlled defined as <140/90 mm Hg by insurance (Commercial, Medicaid, Medicare, Other and None)
Participation in Home Blood Pressure Monitoring (HBPM) | Beginning of the intervention for the relevant wedge up to 48 months participation
  Percentage of participants eligible for home blood pressure monitoring (HBPM) who agree to participate in HBPM based on EHR documentation
Transmission of home blood pressure readings | First three months following each participant's enrollment in HBPM
  Percentage of participants who participate in HPBM who transmit a least 10 BP readings per month
Chronic disease self-management capacity (QICA) | Pre-intervention and six months post-intervention
  Change in Quality Improvement Capacity Assessment QICA scores, scale range 20-200 with higher indicating better outcomes.
Sustained blood pressure control | Beginning with the 6-month intervention period and up to 48 months participation
  Change in percent of participants with blood pressure in control (<140/90 mm Hg) post-intervention
Cost Analysis | Up to 48 months participation
  Marginal changes in net revenue (marginal billing and bonus revenue) and marginal changes in costs related to time for training, staffing costs, and BP monitor

OTHER OUTCOMES:
Clinician mean blood pressure (BP) goal (mm Hg) for patients | Up to 48 months participation
  We will calculate the mean BP goal for each clinician based on the specified BP goal listed in EHR smartphrase for each of the clinician's patients. The mean goal is calculated by the sum of all systolic (SBP) and diastolic BP (DBP) goals divided by the number of patients with goals for each participating clinician. A reasonable range of mean BP goals are: SBP: 120-150 mm Hg and DBP: 80-100 mm Hg for different clinicians
Anti-hypertensive medication intensification | Up to 48 months participation
  Frequency of anti-hypertensive medication intensification (e.g., the number of additions/deletions of anti-hypertensive medication and/or number of changes in dose of anti-hypertensive medication)
The percentage of participants who are managed by a clinical pharmacist | Up to 48 months participation
  The percentage of HBPM participants who are managed by a clinical pharmacist based on EHR data
Team function | Up to 48 months participation
  Change in team function score based on the score on the TEAMS Tool scale at pre-intervention and post-intervention periods for that wedge. Scale range 14-70 with higher scores indicating better outcomes.
Exploratory outcomes- LDL control levels | Up to 48 months participation
  Change in LDL-cholesterol level (mg/dl) based on lipid blood testing in the EHR over 48 months.
Exploratory outcomes- Smoking status | Up to 48 months participation
  Change in percent of current smokers among eligible participants based on EHR documentation over 48 months.
Exploratory outcomes- Hypertension-related Emergency department visits | Up to 48 months participation
  Change in emergency department visits (number) involving a primary diagnosis of hypertension diagnosis among eligible patients recorded on the emergency department discharge summary from the EHR over 48 months.
Exploratory outcomes- Hypertension-related Hospitalizations | Up to 48 months participation
  Change in hospitalization (number) involving a primary diagnosis of hypertension diagnosis among eligible patients recorded on the hospital discharge summary from the EHR over 48 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Fiscella, MD, MPH, Principal Investigator — URMC
Locations (1):
- Highland Family Medicine, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data Quality and Management
  a. Description of Plan for Data Quality and Management - The PI will review all data collection forms on an ongoing basis for data completeness and accuracy as well as protocol compliance. A statement reflecting the results of the review will be sent to the NIH in the annual report. The EHR is the primary data source. EHR data quality will be assessed using extreme outlier data, missing data for outcome variables (i.e. office or transmitted blood pressure readings, dates of visits, participant ID), and loss to follow-up (no data for the participant appears in EHR, e.g. due to relocation, left practice etc). Note: clinical staff will conduct outreach to all participants as part of sound clinical practice. Regular data checks and data cleaning will be deployed to optimize data quality. Multiple imputation methods will be used as necessary to address missing data as described in the statistical analysis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No personally identifiable information will be transcribed. The de-identified data will be stored in a password-protected file on a secure URMC shared drive housed in the Department of Family Medicine. Only the research team will have access to the de-identified data. 7 years after the completion of the study, the audio recordings will destroyed.
URL: https://www.rochester.edu/orpa/

REFERENCES:
- [Derived] Fiscella KA, Sass E, Sridhar SB, Maguire JA, Lashway K, Wong G, Thien A, Thomas M, Bisognano JD, Rosenberg T, Sanders MR, Johnson BA, Polgreen LA. Team-based home blood pressure monitoring for blood pressure equity a protocol for a stepped wedge cluster randomized trial. Contemp Clin Trials. 2023 Nov;134:107332. doi: 10.1016/j.cct.2023.107332. Epub 2023 Sep 16. PMID 37722482

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT05488795/Prot_SAP_000.pdf